CLINICAL TRIAL: NCT06210100
Title: Efficacy and Safety of Accelerated Intermittent Theta Burst Stimulation on Non-suicidal Self-injury and Suicide Behaviors in Adolescents With Unipolar or Bipolar Depression
Brief Title: aiTBS for NSSI and Suicide in Adolescent Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS20230801
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Non Suicidal Self Injury; Suicidal Ideation; Suicide and Self-harm
Keywords: NSSI; MDD; TMS
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial testing iTBS versus sham
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Active Comparator): Active Intermittent theta burst stimulation to the dorsolateral prefrontal cortex; 5 sessions per day, for 10 days.
  Interventions: Device: Active iTBS
- Sham stimulation (Sham Comparator): Sham stimulation to the dorsolateral prefrontal cortex; 5 sessions per day, for 10 days.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Active iTBS — Mag-TD stimulator
  Arms: Active stimulation
Device: Sham iTBS — Mag-TD stimulator
  Arms: Sham stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has been successfully used to help patients with treatment resistant depression. However, its role in alleviating self injuries with and without suicidal ideation remained uncertain. This trial will compare the effectiveness of active accelerated intermittent theta burst stimulation (aiTBS) rTMS to a placebo control on non-suicidal self injury (NSSI) and suicidal attempts in patients with major depressive disorder.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of aiTBS in depressive patients with NSSI or suicidal thoughts and behaviors by measuring changes in clinical ratings at baseline, after all the treatments, and 4 weeks, 8 weeks after treatment. 60 inpatients will be randomized to receive active or sham interventions administered to the left dorso-lateral prefrontal cortex. The treatment will apply active aiTBS rTMS involving 1800 pulses (9 minutes), 5x daily at 60 minutes intervals for 10 days. Changes in mood from baseline to the end of the study will be measured with The Hamilton Rating Scale for Depression-17 item (HAM-D17), Hamilton Anxiety Scale (HAMA) and Young's Mania Scale (YMRS). Non-suicidal self injury will be assessed by the Deliberate Self-Harm Inventory (DSHI) and the Ottawa self-injury inventory (OSI). Suicidal ideation and behaviors assessments include Beck Suicidal Scale Inventory (BSI), the Columbia-Suicide Severity Rating Scale (C-SSRS), and several questions from Self-Injurious Thoughts and Behaviors Interview - Revised (SITBI-R). The World Health Organization Disability Assessment Schedule for children (WHODAS-Child) will be used to evaluate the overall function of adolescent patients. Treatment Emergent Symptom Scale (TESS) would be used to eliminate side effects of combined drugs at baseline and the adverse event record form (AERF) will be used to appraise the safety of aiTBS treatment using these parameters. Changes of brain structure and brain activities will be acquired by pre and post-interventional magnetic resonance imaging (MRI). Fasting blood exams will be conducted to measuring the level of NSSI related endocrine and metabolic changes. To record the change in sensitivity to pain and examine the tolerability of the treatment for these participants, visual analogue scale (VAS) is employed after completing 5 sessions treatment every day.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders 5th Edition) diagnostic criteria for major depressive disorder.
2. Patients aged 12-18 years with at least one guardian to monitor them for 3 months
3. HAMD-17 Total score ≥18
4. Hospitalized patients who had two or more non-suicidal self-injury behaviors meeting the DSM-5 diagnostic criteria in the week before admission (NSSI behavior of more than 5 days in the past year, and a baseline DSHI score ≥2 )
5. Obtain informed consent from patients and guardians

Exclusion Criteria:

1. Substance abusers such as psychoactive drugs or alcohol.
2. Severe physical disability and unable to complete follow-up.
3. Comorbid other major mental illnesses that meet the DSM-5 criteria, such as bipolar disorder, schizophrenia, mental retardation, dementia, severe cognitive impairment, attention deficit hyperactivity disorder, etc.
4. Suffering from any severe physical disease, neurological disease, traumatic brain injury, etc, that affects the structure or function of the brain in the lifetime.
5. Unable to read, understand and complete the assessment or to cooperate with the investigators.
6. Any implants covering a pacemaker, metallic or magnetic objects in the body, or other conditions not suitable for rTMS.
7. A history or family history of epilepsy and other contraindications to TMS.
8. Daily use of benzodiazepines (more than 2mg/d), theophylline, stimulants such as methylphenidate, anticonvulsants, etc.
9. Those who have received systematic psychotherapy (interpersonal relationship therapy, dynamic therapy, cognitive behavioral therapy) or TMS within 3 months before baseline.
10. Other examination abnormalities considered to be inappropriate by investigators.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Deliberate Self-Harm Inventory (DSHI) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Containing one subscale ranging from 0 to 57 to measure the frequencies of NSSI behavior and one subscale ranging from 0 to 76 to measure the severity of NSSI behavior.

SECONDARY OUTCOMES:
Changes in Hamilton Anxiety Scale (HAMA) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Range from 0-56, higher score indicates more severe symptoms
Changes in the 17-item Hamilton Rating Scale for Depression (HAMD-17) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Range from 0-52, higher score indicates more severe symptoms
Changes in Young's Mania Scale (YMRS) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Range from 0-60, higher score indicates more severe symptoms
Changes in Beck Suicidal Scale Inventory (BSI) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Range from 0- 38, higher score indicates more severe suicide ideation.
Changes in The Clinical Global Impression (CGI) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Containing two subscales ranging from 1 to 7 each to measure the symptom severity and overall improvement respectively. Higher score indicates greater severity or greater improvements.
Changes in the subscale of addiction of NSSI from OSI (Ottawa self-injury inventory) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Range from 0- 28, higher score indicates higher addiction.
Changes in the Deliberate Self-Harm Inventory-ideation (DSHI-ideation) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  Range from 0 to 57 to measure the frequency of NSSI ideation
Changes in the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, next day after 10 treatment days, 4 week and 8 week post-treatment
  The C-SSRS is made up of ten categories, all of which maintain binary responses (yes/no) to indicate a presence or absence of the behavior. The ten categories included in the C-SSRS are as follows: Category 1 - Wish to be Dead; Category 2 - Non-specific Active Suicidal Thoughts; Category 3 - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Category 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Category 5 - Active Suicidal Ideation with Specific Plan and Intent; Category 6 - Preparatory Acts or Behavior; Category 7 - Aborted Attempt; Category 8 - Interrupted Attempt; Category 9 - Actual Attempt (non-fatal); Category 10 - Completed Suicide.
  A yes/no binary response is also utilized in assessing self-injurious behavior without suicidal intent. The outcome of the C-SSRS is a numerical score obtained from the aforementioned categories.
Changes in the The World Health Organization Disability Assessment Schedule for children (WHODAS2-child) | Baseline, 4 week and 8 week post-treatment
  The WHODAS-Child is a self-report assessment of difficulties in six domains: understanding and communicating ranging from 0 to 24, getting around ranging from 0 to 20, self-care ranging from 0 to 16, getting along with people ranging from 0 to 20, life activities ranging from 0 to 36, and participation in society ranging from 0 to 20. Higher score indicates worse global function.
Changes of high-resolution T1-weighted anatomical images | Baseline, next day after 10 treatment days, and 8 week post-treatment
  Resting-state MRI (rs-MRI) will be used to exam the change of brain structure. T1-weighted images will be acquired using 3D inversion recovery-prepared fast spoiled gradient-echo sequences.
Changes of Diffusion Tensor Imaging | Baseline, next day after 10 treatment days, and 8 week post-treatment
  Resting-state MRI (rs-MRI) will be used to exam the change of brain structure. Diffusion Tensor Imaging (DTI) will be performed using diffusion-weighted echo planar imaging sequences.
Changes of blood oxygenation level dependent (BOLD) functional imaging signals | Baseline, next day after 10 treatment days, and 8 week post-treatment
  Functional MRI (fMRI) will be used to exam the change of brain function.
Changes in plasma β-endorphin | Baseline, next day after 10 treatment days, and 8 week post-treatment
  in ng/ml
Changes in plasma cortisol | Baseline, next day after 10 treatment days, and 8 week post-treatment
  in ng/ml
Changes in serum Brain-derived neurotrophic factor (BDNF) | Baseline, next day after 10 treatment days, and 8 week post-treatment
  in ng/ml

OTHER OUTCOMES:
Borderline features of patients with NSSI | Baseline
  Measured by The Borderline Personality Feature Scale for Children-11 (BPFS-C-11) ranging from 24 to 120. Higher score indicates stronger borderline personality tendency.
Child maltreatment of patients with NSSI | Baseline
  Measured by the Childhood Trauma Questionnaire (CTQ) ranging from 25 to 125. Higher score indicates more adversity experienced in childhood.
Fundamental parental style of caregivers of patients with NSSI | Baseline
  Measured by the Parental Bonding Instrument (PBI) containing two subscales ranging from 0 to 75 for both mother and father version. Each subscale include 25 item questions, including 12 'care' items and 13 'overprotection' items. For mothers, a care score of 27.0 indicates higher care and a protection score of 13.5 indicates high protection. For fathers, a care score of 24.0 indicates high care and a protection score of 12.5 indicates high protection. high and low categories of care and protection can be combined into four parental bonding types of affectionate constraint, affectionless control, optimal parenting, and neglectful parenting.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline
  Recording any side effects in the adverse event record form (AERF).
Peer relationship of patients with NSSI | Baseline
  Measured by the Peer relationship questionnaire (PRQ) containing 22 items scoring from 22 to 88. The higher the scores on the questionnaire indicate the worse the peer relationships.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second People's Hospital of Dali Bai Autonomous Prefecture, Dali, Yunnan
  - Mental Health Institute of Second Xiangya Hospital, Changsha